CLINICAL TRIAL: NCT02210221
Title: Collaborative European NeuroTrauma Effectiveness Research in TBI (CENTER-TBI)
Brief Title: CENTER-TBI: Collaborative European NeuroTrauma Effectiveness Research in TBI
Acronym: CENTER-TBI
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: University of Cambridge (Other); Erasmus Medical Center (Other); San Gerardo Hospital (Other); University of Sheffield (Other); University of California, San Francisco (Other); Karolinska Institutet (Other); ICON plc (Industry); GABO:mi (Industry); icometrix (Industry)
Responsible Party: Principal Investigator, Andrew Maas, M.D., PhD, Project Coordinator CENTER-TBI, University Hospital, Antwerp
Other Study IDs: 602150
Record Dates: First submitted 2014-07-29; First posted 2014-08-06 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-04

CONDITIONS: Traumatic Brain Injury
Keywords: TBI
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — whole blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The research aims of the CENTER-TBI study are to:

1. better characterize Traumatic Brain Injury (TBI) as a disease and describe it in a European context, and
2. identify the most effective clinical interventions for managing TBI.

Specific aims

1. To collect high quality clinical and epidemiological data with repositories for neuro-imaging, DNA, and serum from patients with TBI.
2. To refine and improve outcome assessment and develop health utility indices for TBI.
3. To develop multidimensional approaches to characterisation and prediction of TBI.
4. To define patient profiles which predict efficacy of specific interventions ("Precision Medicine").
5. To develop performance indicators for quality assurance and quality improvement in TBI care.
6. To validate the common data elements (CDEs) for broader use in international settings, and to develop a user-friendly web based data entry instrument and case report form builder.
7. To develop an open database compatible with Federal Interagency Traumatic Brain Injury Research (FITBIR).
8. To intensify networking activities and international collaborations in TBI.
9. To disseminate study results and management recommendations for TBI to health care professionals, policy makers and consumers, aiming to improve health care for TBI at individual and population levels.
10. To develop a "knowledge commons" for TBI, integrating CENTER-TBI outputs into systematic reviews.

DETAILED DESCRIPTION:
• Introduction:

CENTER-TBI (Collaborative European NeuroTrauma Effectiveness Research in TBI) (www.center-tbi.eu) is a project embedded within the International Initiative on TBI Research (InTBIR) (http://intbir.nih.gov/), as a collaboration between the European Commission (EC), the US National Institute of Neurological Disorders and Stroke (NIH-NINDS) and the Canadian Institute of Health Research (CIHR).

* Research aims:

The basic concept of this project is to exploit the existing heterogeneity in biology, care and outcome of TBI patients to discover underlying pathophysiology, to refine characterisation, and to identify effective clinical interventions. The key driver of our research plan is to collect data from a large number of European centres and sufficiently large cohort to enable 'Comparative effectiveness research' (CER) analyses of differences in clinical care and management pathways in TBI.

Improved disease characterization will aid Precision Medicine, a concept recently enunciated by the US National Academy of Science. Such improved characterization and stratification will allow for more targeted therapies. Further, CER provides a promising framework to identify best practices and improve outcome after TBI. CER is the generation and synthesis of evidence that compares the benefits and harms of alternative methods to prevent, diagnose, treat, and monitor a clinical condition or to improve the delivery of care. The purpose of CER is to assist consumers, clinicians, purchasers, and policy makers to make informed decisions that will improve health care at both the individual and population levels.

* Cohort:

A large core cohort of patients across the severity spectrum in TBI will be recruited at approximately 77 sites in Europe and Israel (the CENTER-TBI Core Study): 5400 patients differentiated into 3 equal strata of approximately 1800:

* ER stratum: patients seen and discharged from the ER;
* Admission stratum: patients admitted to the hospital but not to the ICU;
* ICU stratum: patients admitted directly to the ICU. Balance in numbers between the strata will be aimed for, but sites will be allowed to arrange recruitment strategies to best suit their local requirements.

The core cohort will be underpinned by comparison with a larger registry (the CENTER-TBI registry) based on pragmatic data collection of all patients with TBI seen in participating centres (to establish the internal generalizability of our study), and by comparison with national trauma registries (to establish the external generalizability of our findings).

In the core cohort, detailed data will be collected on clinical parameters, neuroimaging studies, biomarker analyses, DNA analyses, and longitudinal outcome assessments. In selected centres, extended studies will additionally focus on advanced magnetic resonance (MR) imaging, detailed coagulation profiling and high resolution ICU monitoring.

* Sample size assessment:

The sample size estimate (n=5400) was based on:

* Practical logistic considerations
* Power calculations for the different strata, targeting comparative effectiveness analyses, assuming a between-centre and between-country heterogeneity as identified in previous research (expressed by variance parameter from a random effects model, Tau^2 of 0.431)
* Postulated odds ratios for intervention effects of approximately 5% improvement in outcome.

Overall, these calculations provided a statistical power to detect odds ratios of ~1.2 associated with differences in process or intervention variables across the core dataset with a power of 80%; and require somewhat larger odds ratios in each of the three individual strata. In the registry we expect to be able to detect differences (predominantly in organizational or system variables) with an odds ratio of 1.2 with a power of 82%.

* Quality control and assurance:

Continuous monitoring of enrolment and completeness of data will be performed by ICON as contract research organization (CRO). Source data verification (SDV) will be performed in 10% of subjects by the CRO. The quality of data collection will be further enhanced by implementing automated data entry checks for impossible/implausible values and implementing data checks for consistency between variables. A task force of study personnel will evaluate the completeness, consistency and validity of submitted data and function as support desk for participating sites.

* Data management:

Prior to upload to the study database, all acquired data will be stored locally. All patients will be allocated a random Global Unique Personal Identification number (GUPI) which will be linked locally to hospital identifiers. All uploaded data will be de-identified and images will be defaced prior to upload. While blood samples and clinical data will be linked, both sets of data will be kept confidential and anonymised beyond the initial stage of correlation for analysis. All imaging and electronic data will be kept on individually password protected servers. All clinical data will be entered into electronic Case Report Forms (eCRFs) and managed by the 'QuesGen data management platform' (http://www.quesgen.com/) which will be developed in collaboration with Karolinska Institutet International Neuroinformatics Coordinating Faculty (KI-INCF). As data is entered into each form, the system will run data validation checks that include conditionally required data, validation across fields, and validation requirements based on subject type. If any validation check fails, the user is alerted immediately that the data does not meet Quality Assurance (QA) criteria and the issue can be addressed and corrected at that point. All de-identified electronic study data in the CENTER-TBI database will be stored securely in the European data space under supervision of KI-INCF for the duration of subject enrolment and follow-up and for a period afterwards for data analysis and preparation of publications. We estimate that the analysis and publication period will last for several years after the conclusion of subject enrolment.

Together with QuesGen Systems, KI-INCF will ensure that data standards are established for the data model e.g. conformity of field formats, field codes and names to ensure consistency across all datasets. Any approved changes will be fully documented with dataset updates to maintain data quality and accuracy. KI-INCF will be responsible for importing cleaned datasets to other analytic platforms as determined by the coordinators.

Where applicable, information relevant to the patient's care will be made available to the physician responsible. Data, including blood samples collected as part of this study will be shared in an anonymised form with collaborators from other European states (this is part of a European Commission Framework7 funded program), and with selected collaborators in other countries who form part of an emerging International Traumatic Brain Injury Research initiative.

* Computing platform and Neuroinformatics Resource:

The KI-INCF will coordinate the establishment of an informatics platform for acquisition, storage and analysis of CDE-based clinical data. The goal is to develop a next generation open standards-based platform to support advanced large-scale analytics and model building. Such a platform also provides a model for future clinical studies on brain diseases and disorders. This development will receive additional support from One Mind for Research.

* Statistical analysis plan:

Statistical analyses for the Comparative Effectiveness Research (CER) questions will primarily apply random effects modelling, in which center is included at the higher level, and patients are considered clustered within centers. In some analyses, higher levels of clustering will also be considered, e.g. country, or European region; or lower levels, e.g. physicians within hospitals. Confounding factors as measured at the individual patient and/or center level, will be considered extensively, and will be targeted to the specific research question.

Statistical analyses for better characterization of TBI will be exploratory, aiming to better understand the complexity of the disease and to discover new associations. In addition to standard statistical descriptive and inferential techniques, we will also employ novel machine learning techniques as appropriate.

Prognostic analyses will consider a range of variables, including genetic, demographic and clinical data, physiological signals, imaging results, and biomarkers as predictors of early endpoints and physiologic derangement (e.g. raised ICP), and late outcome, including mortality, functional outcome, quality of life and neuropsychological performance. Previously and newly developed prediction models will be validated by comparison of observed to predicted outcome risks, with predictive performance summarized by measures for model fit, discrimination, and calibration.

* Missing data:

Every effort will be made to limit the number of missing data in the CENTER-TBI study. Missing values are, however, inherent to any clinical study. Missing values may confound the descriptive, prognostic and CER analyses. Thus, appropriate techniques for dealing with missing values are required. First, we will evaluate the various reasons for missingness per centre. Next, we will explore the use of alternative statistical approaches, including inverse probability weighting and multiple imputation. We will consider missing values in baseline characteristics as well as in short and long term outcomes. Based on simulation studies and practical considerations we will develop standard operating procedures towards the analyses with missing values, respecting the differences in multiple research questions.

* Informed Consent:

Informed consent procedures will follow local and national requirements in all cases. We anticipate that many potential patients will not be able to consent themselves to participate in this project. The nature of TBI means that some patients may lack capacity to decide to participate in this study especially at the earliest time point. It is important to try and include these patients to ensure that representative samples of patients are included to avoid bias in the study findings. Every step will be taken to ensure that a test of capacity is undertaken before a decision on a person's capacity to consent or not to consent to participation in research is taken. If the subject is not capable of self-consent, all efforts will be made to locate a legally acceptable representative to act on behalf of the subject. When a legally acceptable representative (e.g. consultee/proxy) is identified, their opinion will be sought about the potential participant's wishes and feelings in relation to the project, and whether he or she would have wanted to take part in the study.

Subjects are free to withdraw, or be withdrawn by their consultee/proxy if appropriate, at any point in the study, and they need not state a reason.

* Impact:

The CENTER-TBI project will contribute towards the overall goals of InTBIR, by identifying more effective and efficient treatment provision, thus improving outcome and reducing costs. The science in the project will provide novel information on disease processes, treatment, outcome, and prognosis in TBI, identifying new therapeutic targets and therapies; while the CENTER-TBI repositories will ensure opportunities for legacy research. Thus, the project has the potential to improve current health care and its delivery at both population and individual levels, deliver early scientific advances that could improve the care of patients with TBI, and provide a rich investment for future biomedical research.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of TBI
* Clinical indication for CT scan
* Presentation within 24 hours of injury
* Informed consent obtained according to local and national requirements

Exclusion Criteria:

* Severe pre-existing neurological disorder that would confound outcome assessments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting with traumatic brain injury.
  The data collection will be stratified upon enrolment into 3 clinical groups differentiated by clinical care path:
  * ER stratum: patients seen and discharged from the ER
  * Admission stratum: patients admitted to hospital but not to the ICU
  * ICU stratum: patients admitted directly to the ICU
Sampling Method: Non-Probability Sample
Enrollment: 4559 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Maas, MD, PhD, Study Chair — Antwerp University Hospital / University of Antwerp, Edegem, Belgium; David Menon, MD, PhD, Study Director — University of Cambridge, Addenbrookes hospital, Cambridge, UK
Locations (65):
- Austria (2):
  - Innsbruck Medical University, Innsbruck
  - Medical University Vienna, Vienna
- Belgium (4):
  - Antwerp University Hospital, Edegem
  - University Hospitals Leuven, Leuven
  - CHR Citadelle, Liège
  - CHU Liege, Liège
- Denmark (2):
  - Region Hovedstaden Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Turku University Hospital, Turku
- France (5):
  - University Hospital of Grenoble, Grenoble
  - Lille University Hospital, Lille
  - University Hospital Nancy, Nancy
  - APHP, Paris
  - CHU Poitiers, Poitiers
- Germany (4):
  - University Hospital Aachen, Aachen
  - Charité Campus Virchow, Berlin
  - University Hospital Heidelberg, Heidelberg
  - Klinikum Ludwigsburg, Ludwigsburg
- Hungary (2):
  - University of Pecs, Pécs
  - University of Szeged, Szeged
- Israel (2):
  - Rambam Medical Center, Haifa
  - Hadassah-hebrew University Medical Center, Jerusalem
- Italy (8):
  - Bufalini Hospital, Cesena
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Poloclinico, Milan
  - Niguarda Hospital, Milan
  - S Raffaele University Hospital, Milan
  - ASST di Monza, Monza
  - Maggiore Della Carità Hospital, Novara
  - Azienda Ospedaliera Università di Padova, Padua
  - AOU Città della Salute e della Scienza di Torino, Torino
- Latvia (3):
  - Rezekne Hospital, Rēzekne
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga Eastern Clinical University Hospital, Riga
- Lithuania (3):
  - University of Health Sciences, Kaunas
  - Center of neurovascular surgery, Clinic of neurology and neurosurgery, Vilnius University, Vilnius
  - Kaunas University of technology and Vilnius University, Vilnius
- Netherlands (7):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Radboud University Medical Center, Nijmegen
  - Erasmus MC, Rotterdam
  - Medical Center Haaglanden, The Hague
  - The HAGA Hospital, The Hague
  - TweeSteden Ziekenhuis, Tilburg
- Norway (3):
  - Oslo University Hospital, Oslo
  - University Hospital Northern Norway, Tromsø
  - St Olavs Hospital/Norwegian University of science and technology, Trondheim
- Emergency County Hospital Timisoara, Timișoara, Romania
- Clinical centre of Vojvodina, Novi Sad, Serbia
- Spain (4):
  - Vall d'Hebron University Hospital, Barcelona
  - Cruces University Hospital, Bilbao
  - Hospital Universitario 12 de Octubre, Madrid
  - Clínico Universitario de Valencia, Valencia
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Umea University Hospital, Umeå
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (9):
  - Queen Elizabeth Hospital, Birmingham
  - Southmead Hospital, Bristol
  - Addenbrookes Hospital, Cambridge
  - Lothian Health Board, Edinburgh
  - The Walton centre NHS Foundation Trust, Liverpool
  - Kings college London, London
  - Salford Royal Hospital, Salford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospitals Southampton NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Jacob L, Castro J, Heslot C, Andelic N, Tenovuo O; CENTER-TBI Participants and Investigators (Appendix); Azouvi P. Absence from work in the 12 months following mild traumatic brain injury in Europe: a CENTER-TBI cohort study. Ann Phys Rehabil Med. 2025 Nov;68(8):102017. doi: 10.1016/j.rehab.2025.102017. Epub 2025 Sep 30. PMID 41032948
- [Derived] Kals M, Wilson L, Levey DF, Parodi L, Steyerberg EW, Richardson S, He F, Sun X, Jain S, Palotie A, Ripatti S, Rosand J, Manley GT, Maas AIR, Stein MB, Menon DK; Genetic Associations In Neurotrauma (GAIN) Consortium (with contribution from the CENTER-TBI and TRACK-TBI studies). Genetic vulnerability and adverse mental health outcomes following mild traumatic brain injury: a meta-analysis of CENTER-TBI and TRACK-TBI cohorts. EClinicalMedicine. 2024 Dec 5;78:102956. doi: 10.1016/j.eclinm.2024.102956. eCollection 2024 Dec. PMID 39720422
- [Derived] Guglielmi A, Graziano F, Bogossian EG, Turgeon AF, Taccone FS, Citerio G; CENTER-TBI Participants and Investigators. Haemoglobin values, transfusion practices, and long-term outcomes in critically ill patients with traumatic brain injury: a secondary analysis of CENTER-TBI. Crit Care. 2024 Jun 14;28(1):199. doi: 10.1186/s13054-024-04980-6. PMID 38877571
- [Derived] Pisica D, Volovici V, Yue JK, van Essen TA, den Boogert HF, Vande Vyvere T, Haitsma I, Nieboer D, Markowitz AJ, Yuh EL, Steyerberg EW, Peul WC, Dirven CMF, Menon DK, Manley GT, Maas AIR, Lingsma HF; CENTER-TBI Participants and Investigators. Clinical and Imaging Characteristics, Care Pathways, and Outcomes of Traumatic Epidural Hematomas: A Collaborative European NeuroTrauma Effectiveness Research in Traumatic Brain Injury Study. Neurosurgery. 2024 Nov 1;95(5):986-999. doi: 10.1227/neu.0000000000002982. Epub 2024 May 21. PMID 38771081
- [Derived] Vreeburg RJG, Singh RD, van Erp IAM, Korhonen TK, Yue JK, Mee H, Timofeev I, Kolias A, Helmy A, Depreitere B, Moojen WA, Younsi A, Hutchinson P, Manley GT, Steyerberg EW, de Ruiter GCW, Maas AIR, Peul WC, van Dijck JTJM, den Boogert HF, Posti JP, van Essen TA; for the CENTER-TBI Participants and Investigators. Early versus delayed cranioplasty after decompressive craniectomy in traumatic brain injury: a multicenter observational study within CENTER-TBI and Net-QuRe. J Neurosurg. 2024 Apr 26;141(4):895-907. doi: 10.3171/2024.1.JNS232172. Print 2024 Oct 1. PMID 38669706
- [Derived] Howe EI, Andelic N, Brunborg C, Zeldovich M, Helseth E, Skandsen T, Olsen A, Fure SCR, Theadom A, Rauen K, Madsen BA, Jacobs B, van der Naalt J, Tartaglia MC, Einarsen CE, Storvig G, Tronvik E, Tverdal C, von Steinbuchel N, Roe C, Hellstrom T; CENTER-TBI Participants and Investigators. Frequency and predictors of headache in the first 12 months after traumatic brain injury: results from CENTER-TBI. J Headache Pain. 2024 Mar 25;25(1):44. doi: 10.1186/s10194-024-01751-0. PMID 38528477
- [Derived] Zeldovich M, Bockhop F, Covic A, Mueller I, Polinder S, Mikolic A, van der Vlegel M, von Steinbuechel N; CENTER-TBI participants and investigators. Factorial validity and comparability of the six translations of the Rivermead Post-Concussion Symptoms Questionnaire translations: results from the CENTER-TBI study. J Patient Rep Outcomes. 2023 Sep 8;7(1):90. doi: 10.1186/s41687-023-00632-5. PMID 37682406
- [Derived] van Essen TA, van Erp IAM, Lingsma HF, Pisica D, Yue JK, Singh RD, van Dijck JTJM, Volovici V, Younsi A, Kolias A, Peppel LD, Heijenbrok-Kal M, Ribbers GM, Menon DK, Hutchinson PJA, Manley GT, Depreitere B, Steyerberg EW, Maas AIR, de Ruiter GCW, Peul WC; CENTER-TBI Investigators and Participants. Comparative effectiveness of decompressive craniectomy versus craniotomy for traumatic acute subdural hematoma (CENTER-TBI): an observational cohort study. EClinicalMedicine. 2023 Aug 9;63:102161. doi: 10.1016/j.eclinm.2023.102161. eCollection 2023 Sep. PMID 37600483
- [Derived] Lang L, Wang T, Xie L, Yang C, Skudder-Hill L, Jiang J, Gao G, Feng J. An independently validated nomogram for individualised estimation of short-term mortality risk among patients with severe traumatic brain injury: a modelling analysis of the CENTER-TBI China Registry Study. EClinicalMedicine. 2023 Apr 28;59:101975. doi: 10.1016/j.eclinm.2023.101975. eCollection 2023 May. PMID 37180469
- [Derived] Howe EI, Zeldovich M, Andelic N, von Steinbuechel N, Fure SCR, Borgen IMH, Forslund MV, Hellstrom T, Soberg HL, Sveen U, Rasmussen M, Kleffelgaard I, Tverdal C, Helseth E, Lovstad M, Lu J, Arango-Lasprilla JC, Tenovuo O, Azouvi P, Dawes H, Roe C; CENTER-TBI participants and investigators. Rehabilitation and outcomes after complicated vs uncomplicated mild TBI: results from the CENTER-TBI study. BMC Health Serv Res. 2022 Dec 16;22(1):1536. doi: 10.1186/s12913-022-08908-0. PMID 36527074
- [Derived] Rezoagli E, Petrosino M, Rebora P, Menon DK, Mondello S, Cooper DJ, Maas AIR, Wiegers EJA, Galimberti S, Citerio G; CENTER-TBI, OzENTER-TBI Participants and Investigators. High arterial oxygen levels and supplemental oxygen administration in traumatic brain injury: insights from CENTER-TBI and OzENTER-TBI. Intensive Care Med. 2022 Dec;48(12):1709-1725. doi: 10.1007/s00134-022-06884-x. Epub 2022 Oct 20. PMID 36264365
- [Derived] Akerlund CAI, Holst A, Stocchetti N, Steyerberg EW, Menon DK, Ercole A, Nelson DW; CENTER-TBI Participants and Investigators. Clustering identifies endotypes of traumatic brain injury in an intensive care cohort: a CENTER-TBI study. Crit Care. 2022 Jul 27;26(1):228. doi: 10.1186/s13054-022-04079-w. PMID 35897070
- [Derived] Volovici V, Pisica D, Gravesteijn BY, Dirven CMF, Steyerberg EW, Ercole A, Stocchetti N, Nelson D, Menon DK, Citerio G, van der Jagt M, Maas AIR, Haitsma IK, Lingsma HF; CENTER-TBI investigators, participants for the ICU stratum. Comparative effectiveness of intracranial hypertension management guided by ventricular versus intraparenchymal pressure monitoring: a CENTER-TBI study. Acta Neurochir (Wien). 2022 Jul;164(7):1693-1705. doi: 10.1007/s00701-022-05257-z. Epub 2022 Jun 1. PMID 35648213
- [Derived] van Essen TA, Lingsma HF, Pisica D, Singh RD, Volovici V, den Boogert HF, Younsi A, Peppel LD, Heijenbrok-Kal MH, Ribbers GM, Walchenbach R, Menon DK, Hutchinson P, Depreitere B, Steyerberg EW, Maas AIR, de Ruiter GCW, Peul WC; CENTER-TBI Collaboration Group. Surgery versus conservative treatment for traumatic acute subdural haematoma: a prospective, multicentre, observational, comparative effectiveness study. Lancet Neurol. 2022 Jul;21(7):620-631. doi: 10.1016/S1474-4422(22)00166-1. Epub 2022 May 5. PMID 35526554
- [Derived] Holthe IL, Dahl HM, Rohrer-Baumgartner N, Eichler S, Elseth MF, Holthe O, Berntsen T, Yeates KO, Andelic N, Lovstad M. Neuropsychological Impairment, Brain Injury Symptoms, and Health-Related Quality of Life After Pediatric TBI in Oslo. Front Neurol. 2022 Jan 28;12:719915. doi: 10.3389/fneur.2021.719915. eCollection 2021. PMID 35153967
- [Derived] Huijben JA, Pisica D, Ceyisakar I, Stocchetti N, Citerio G, Maas AIR, Steyerberg EW, Menon DK, van der Jagt M, Lingsma HF. Pharmaceutical Venous Thrombosis Prophylaxis in Critically Ill Traumatic Brain Injury Patients. Neurotrauma Rep. 2022 Jan 7;2(1):4-14. doi: 10.1089/neur.2021.0037. eCollection 2022. PMID 35112104
- [Derived] Galimberti S, Graziano F, Maas AIR, Isernia G, Lecky F, Jain S, Sun X, Gardner RC, Taylor SR, Markowitz AJ, Manley GT, Valsecchi MG, Bellelli G, Citerio G; CENTER-TBI and TRACK-TBI participants and investigators. Effect of frailty on 6-month outcome after traumatic brain injury: a multicentre cohort study with external validation. Lancet Neurol. 2022 Feb;21(2):153-162. doi: 10.1016/S1474-4422(21)00374-4. PMID 35065038
- [Derived] Puybasset L, Perlbarg V, Unrug J, Cassereau D, Galanaud D, Torkomian G, Battisti V, Lefort M, Velly L, Degos V, Citerio G, Bayen E, Pelegrini-Issac M; MRI-COMA Investigators CENTER-TBI MRI Participants and MRI Only Investigators. Prognostic value of global deep white matter DTI metrics for 1-year outcome prediction in ICU traumatic brain injury patients: an MRI-COMA and CENTER-TBI combined study. Intensive Care Med. 2022 Feb;48(2):201-212. doi: 10.1007/s00134-021-06583-z. Epub 2022 Dec 14. PMID 34904191
- [Derived] Citerio G, Robba C, Rebora P, Petrosino M, Rossi E, Malgeri L, Stocchetti N, Galimberti S, Menon DK; Center-TBI participants and investigators. Management of arterial partial pressure of carbon dioxide in the first week after traumatic brain injury: results from the CENTER-TBI study. Intensive Care Med. 2021 Sep;47(9):961-973. doi: 10.1007/s00134-021-06470-7. Epub 2021 Jul 24. PMID 34302517
- [Derived] Robba C, Rebora P, Meyfroidt G, Citerio G. The authors reply. Crit Care Med. 2021 May 1;49(5):e554-e555. doi: 10.1097/CCM.0000000000004961. No abstract available. PMID 33854024
- [Derived] Huijben JA, Dixit A, Stocchetti N, Maas AIR, Lingsma HF, van der Jagt M, Nelson D, Citerio G, Wilson L, Menon DK, Ercole A; CENTER-TBI investigators and participants. Use and impact of high intensity treatments in patients with traumatic brain injury across Europe: a CENTER-TBI analysis. Crit Care. 2021 Feb 23;25(1):78. doi: 10.1186/s13054-020-03370-y. PMID 33622371
- [Derived] Borgen IMH, Roe C, Brunborg C, Tenovuo O, Azouvi P, Dawes H, Majdan M, Ranta J, Rusnak M, Wiegers EJA, Tverdal C, Jacob L, Cogne M, von Steinbuechel N, Andelic N; CENTER-TBI participants investigators. Care transitions in the first 6months following traumatic brain injury: Lessons from the CENTER-TBI study. Ann Phys Rehabil Med. 2021 Nov;64(6):101458. doi: 10.1016/j.rehab.2020.10.009. Epub 2021 Jul 23. PMID 33246186
- [Derived] Robba C, Banzato E, Rebora P, Iaquaniello C, Huang CY, Wiegers EJA, Meyfroidt G, Citerio G; Collaborative European NeuroTrauma Effectiveness Research in Traumatic Brain Injury (CENTER-TBI) ICU Participants and Investigators. Acute Kidney Injury in Traumatic Brain Injury Patients: Results From the Collaborative European NeuroTrauma Effectiveness Research in Traumatic Brain Injury Study. Crit Care Med. 2021 Jan 1;49(1):112-126. doi: 10.1097/CCM.0000000000004673. PMID 33060506
- [Derived] Gravesteijn BY, Sewalt CA, Nieboer D, Menon DK, Maas A, Lecky F, Klimek M, Lingsma HF; CENTER-TBI collaborators. Tracheal intubation in traumatic brain injury: a multicentre prospective observational study. Br J Anaesth. 2020 Oct;125(4):505-517. doi: 10.1016/j.bja.2020.05.067. Epub 2020 Jul 31. PMID 32747075
- [Derived] Gao G, Wu X, Feng J, Hui J, Mao Q, Lecky F, Lingsma H, Maas AIR, Jiang J; China CENTER-TBI Registry Participants. Clinical characteristics and outcomes in patients with traumatic brain injury in China: a prospective, multicentre, longitudinal, observational study. Lancet Neurol. 2020 Aug;19(8):670-677. doi: 10.1016/S1474-4422(20)30182-4. PMID 32702336
- [Derived] Robba C, Rebora P, Banzato E, Wiegers EJA, Stocchetti N, Menon DK, Citerio G; Collaborative European NeuroTrauma Effectiveness Research in Traumatic Brain Injury Participants and Investigators. Incidence, Risk Factors, and Effects on Outcome of Ventilator-Associated Pneumonia in Patients With Traumatic Brain Injury: Analysis of a Large, Multicenter, Prospective, Observational Longitudinal Study. Chest. 2020 Dec;158(6):2292-2303. doi: 10.1016/j.chest.2020.06.064. Epub 2020 Jul 4. PMID 32634435
- [Derived] Riemann L, Beqiri E, Smielewski P, Czosnyka M, Stocchetti N, Sakowitz O, Zweckberger K, Unterberg A, Younsi A; CENTER-TBI High Resolution ICU (HR ICU) Sub-Study Participants and Investigators. Low-resolution pressure reactivity index and its derived optimal cerebral perfusion pressure in adult traumatic brain injury: a CENTER-TBI study. Crit Care. 2020 May 26;24(1):266. doi: 10.1186/s13054-020-02974-8. PMID 32456684
- [Derived] Gravesteijn BY, Nieboer D, Ercole A, Lingsma HF, Nelson D, van Calster B, Steyerberg EW; CENTER-TBI collaborators. Machine learning algorithms performed no better than regression models for prognostication in traumatic brain injury. J Clin Epidemiol. 2020 Jun;122:95-107. doi: 10.1016/j.jclinepi.2020.03.005. Epub 2020 Mar 20. PMID 32201256
- [Derived] Huijben JA, Wiegers EJA, Ercole A, de Keizer NF, Maas AIR, Steyerberg EW, Citerio G, Wilson L, Polinder S, Nieboer D, Menon D, Lingsma HF, van der Jagt M; CENTER-TBI investigators and participants for the ICU stratum. Quality indicators for patients with traumatic brain injury in European intensive care units: a CENTER-TBI study. Crit Care. 2020 Mar 4;24(1):78. doi: 10.1186/s13054-020-2791-0. PMID 32131882
- [Derived] Van Essen TA, Volovici V, Cnossen MC, Kolias A, Ceyisakar I, Nieboer D, Peppel LD, Heijenbrok-Kal M, Ribbers G, Menon D, Hutchinson P, Depreitere B, de Ruiter GCW, Lingsma HF, Steyerberg EW, Maas AI, Peul WC. Comparative effectiveness of surgery in traumatic acute subdural and intracerebral haematoma: study protocol for a prospective observational study within CENTER-TBI and Net-QuRe. BMJ Open. 2019 Oct 16;9(10):e033513. doi: 10.1136/bmjopen-2019-033513. PMID 31619435
- [Derived] Steyerberg EW, Wiegers E, Sewalt C, Buki A, Citerio G, De Keyser V, Ercole A, Kunzmann K, Lanyon L, Lecky F, Lingsma H, Manley G, Nelson D, Peul W, Stocchetti N, von Steinbuchel N, Vande Vyvere T, Verheyden J, Wilson L, Maas AIR, Menon DK; CENTER-TBI Participants and Investigators. Case-mix, care pathways, and outcomes in patients with traumatic brain injury in CENTER-TBI: a European prospective, multicentre, longitudinal, cohort study. Lancet Neurol. 2019 Oct;18(10):923-934. doi: 10.1016/S1474-4422(19)30232-7. PMID 31526754
- [Derived] Maas AI, Menon DK, Steyerberg EW, Citerio G, Lecky F, Manley GT, Hill S, Legrand V, Sorgner A; CENTER-TBI Participants and Investigators. Collaborative European NeuroTrauma Effectiveness Research in Traumatic Brain Injury (CENTER-TBI): a prospective longitudinal observational study. Neurosurgery. 2015 Jan;76(1):67-80. doi: 10.1227/NEU.0000000000000575. PMID 25525693
- See also: CENTER - TBI website — https://www.center-tbi.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: CENTER-TBI is an observational cohort study. Data from 4509 patients from 18 countries, collected between Dec 9, 2014, and Dec 17, 2017, are analysed in the core study: 848 (19%) patients were in the ER stratum, 1523 (34%) in the admission stratum, and 2138 (47%) in the ICU stratum.
Pre-assignment Details: Of 4559 patients in the core study, 4509 patients are available for analysis.
Groups:
- CENTER-TBI Population: Data from 4509 patients from 18 countries, collected between Dec 9, 2014, and Dec 17, 2017, were analysed in the core study and from 22 782 patients in the registry. In the core study, 848 (19%) patients were in the ER stratum, 1523 (34%) in the admission stratum, and 2138 (47%) in the ICU stratum.
Period: Overall Study
Arm/Group | CENTER-TBI Population
Started | 4559
Completed | 4509
Not Completed | 50
Not completed — Lack of Efficacy | 7
Not completed — Withdrawal by Subject | 43

BASELINE CHARACTERISTICS:
Groups:
- CENTER-TBI Population: Data from 4509 patients from 18 countries, collected between Dec 9, 2014, and Dec 17, 2017, were analysed in the core study.
Arm/Group | CENTER-TBI Population
Number analyzed (Participants) | 4509
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [30 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1486
  Male | 3023
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Europe | 4509

OUTCOME MEASURES:

1. Primary Outcome: Glasgow Outcome Scale - Extended (GOSE) at 6 Months
Description: The Extended Glasgow Outcome Scale is a global scale for functional outcome that rates patient status into 8 categories, going from dead to good recovery.
  1. Death
  2. Vegetative sate
  3. Lower severe disability
  4. Upper severe disability
  5. Lower moderate disability
  6. Upper moderate disability - some disability but can potentially return to some form of employment
  7. Lower good recovery - minor physical or mental defect
  8. Upper good recovery - full recovery
  The 6-month GOSE score is available in 3804 patients (84%).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- ER Stratum: patients admitted to the ER
- Admission Stratum: patients admitted but not to the ICU
- ICU Stratum: patients admitted to the ICU
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 3804 | 694 | 1264 | 1846
Participants
  6-month GOSE <8 | 2419 | 207 | 665 | 1547
  6-month unfavourable outcome (GOSE <5) | 966 | 31 | 140 | 795
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum in 6-month mortality; Test type: Non-Inferiority — non-inferiority margin = 0; p < 0.0001, ANOVA — No corrections for multiple comparisons were done
Statistical Analysis 2: Comparison: CENTER-TBI Population; Test type: Other; observed to expected ratio = 0.70, 95% CI 2-sided [0.62 to 0.76] — numerator: 6-month mortality observed denominator: 6-month mortality expected 95% CIs estimated according to a Poisson distribution

2. Primary Outcome: SF-12v2 Health Survey (Short-Form Health Survey With 12 Questions) at 6 Months
Description: The SF-12v2 Health Survey uses 12 questions to measure functional health and well-being from the patient's point of view. The SF-12v2 at 6 months is available in 2300 patients.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- ER Stratum: patients in the ER
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 2300 | 480 | 857 | 963
Participants
  6-month SF-12v2 mental component summary <40 (impaired) | 551 | 101 | 184 | 266
  6-month SF-12v2 physical component summary <40 (impaired) | 661 | 112 | 207 | 342
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum in SF-12v2 mental component summary; Test type: Non-Inferiority — non-inferiority margin = 0; p < 0.0001, ANOVA — No corrections for multiple comparisons were done
Statistical Analysis 2: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum in SF-12v2 physical component summary; Test type: Non-Inferiority — non-inferiority margin = 0; p < 0.0001, ANOVA — No corrections for multiple comparisons were done

3. Primary Outcome: 6 Month Quality of Life in Brain Injury (Qolibri-OS) <52 (Impaired)
Description: The Quality of Life in Brain Injury (Qolibri-OS) is a 6 item overall scale that provides a profile of health-related quality of life in domains typicality affected by brain injury, such as physical function, cognition, emotional status, ability to perform daily activities, personal life and social relationship, and satisfaction with current situation and future prospects.
  The QOLIBRI scores are reported on a 0-100 scale , where 0=worst possible quality of life and 100=best possible quality of life.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- ER Stratum: patients at the ER
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 2323 | 474 | 866 | 983
Participants | 511 | 91 | 160 | 260
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum in Qolibri Overall Scale; Test type: Non-Inferiority — non-inferiority margin = 0; p < 0.0001, ANOVA — No corrections for multiple comparisons were done

4. Secondary Outcome: 6 Month Post-traumatic Stress Disorder (PTSD) Checklist for DSM-5 (PCL-5) <33 (Impaired)
Description: The PCL-5 is a self-report rating scale intended to assess 20 DSM-5 symptoms of Posttraumatic Stress Disorder. The standard recall period for the PCL-5 is one month. For CENTER-TBI a recall period of one week was used at the 2-3 week assessment, and the standard one month recall period was used at other time points. The sum of scores can range from 0 to 80, where high scores indicate more pronounced PTSD symptoms.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 2173 | 456 | 818 | 899
Participants | 201 | 40 | 77 | 84
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p < 0.0001, ANOVA — No correlations for multiple comparisons were done

5. Secondary Outcome: 6 Month Rivermead Post Concussion Questionnaire <16 (Impaired)
Description: The Rivermead PCS Questionnaire (RPQ) was originally developed as a measure of severity of symptoms following MTBI. It consists of 16 post-concussion symptoms including headaches, dizziness, nausea/vomiting, noise sensitivity, sleep disturbance, fatigue, irritability, feeling depressed/tearful, feeling frustrated/ impatient, forgetfulness, poor concentration, taking longer to think, blurred vision, light sensitivity, double vision and restlessness. In the original version of the RPQ, participants are asked to rate the degree (on a scale of 0 to 4) to which a particular symptom has been absent or a mild, moderate or severe problem over the previous 7 days compared with premorbid levels. Total scores range from 0 to 64 with higher scores indicating more severe symptoms. Scores equal to or greater than 16 were considered indicative of persisting post-concussion symptoms.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 2259 | 467 | 852 | 940
Participants | 643 | 98 | 200 | 345
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p < 0.0001, ANOVA — No correlations for multiple comparisons were done

6. Secondary Outcome: 6 Month Galveston Orientation and Amnesia Test (GOAT) < 75 (Impaired)
Description: The GOAT is a standardised assessment used to determine whether a participant is in post-traumatic amnesia (PTA). PTA is an early phase of TBI recovery during which the person with injury shows markedly impaired memory, confusion, fluctuation in performance, disorientation, and other neurobehavioral signs and symptoms. GOAT questions assess orientation, memory for the first event that the participant can recall after the injury, and memory for the last event that the participant can recall from before the injury.
  The GOAT's total score must be achieved by subtracting from 100 the total amount of error scores (Total score = 100 - total amount of error scores). Scores lower than 75 point to the fact that the victim is still experiencing amnesia.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 1607 | 281 | 610 | 716
Participants | 67 | 6 | 8 | 53
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p < 0.0001, ANOVA — No correlations for multiple comparisons were done

7. Secondary Outcome: 6 Month Rey Auditory Verbal Learning Test (RAVLT) - Impaired
Description: The Rey Auditory Verbal Learning Test (RAVLT) is a test of verbal memory that assesses the ability to acquire 15 words. Recall is assessed after each presentation of the list, after the recall of an interference list, and again following a 20-minute delay. The total score for recall of the principal list ranges from 0 to 75, with higher scores indicating better performance.
  Impairment was defined as performance that was 1.33 SDs below the mean of a reference group of healthy peers.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 1823 | 368 | 705 | 750
Participants | 350 | 45 | 107 | 198
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p < 0.0001, ANOVA

8. Secondary Outcome: 6 Month Timed up and go Test - Impaired
Description: In the timed up and go (TUG) test, subjects are asked to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again, for quantifying functional mobility. The presence of slowness, hesitancy, abnormal trunk or arm movements, staggering or stumbling is used to grade the patient from 1 (normal) to 5 (severely abnormal). Impaired mobility was defined as taking 14 seconds or longer to perform the TUG test.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 1481 | 293 | 554 | 634
Participants | 342 | 62 | 108 | 172
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p = 0.169, ANOVA

9. Secondary Outcome: 6 Month JK Coma Recovery Scale - Revised <23 (Impaired)
Description: The Coma Recovery Scale- Revised (CRS-R) is a standardized behavioral assessment instrument designed to measure neurobehavioral function in patients with disorders of consciousness (DOC). The CRS-R is comprised of six subscales addressing auditory, visual, motor, oromotor/verbal, communication and arousal functions. Subscale items are hierarchically-arranged, corresponding to brain stem, subcortical and cortically-mediated functions. Scores range between 0 (deep coma) and 23 (able to follow commands and to use objects purposefully). A total score less than 23 indicates impairment.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- ER/Admission Stratum: patients at the ER or patients admitted to hospital but not to the ICU
Arm/Group | CENTER-TBI Population | ER/Admission Stratum | ICU Stratum
Number analyzed (Participants) | 227 | 92 | 135
Participants | 17 | 0 | 17
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p < 0.0001, Fisher Exact

10. Secondary Outcome: 6 Month Trail Making Test (TMT) Part A - Impaired
Description: The Trail Making Test (TMT) is a measure of attention, speed, and mental flexibility. Part A requires the individual to draw lines to connect 25 encircled numbers distributed on a page. Part B is similar except the person must alternate between numbers and letters and is more difficult and takes longer to complete. Both sections are timed and the score represents the amount of time required to complete the task, with shorter times indicating better performance. The maximum time allowed is 100 seconds.
  Impairment cutoff: > 55.9 (based on the comparison group as a whole and expressed as raw score).
  For all the cognitive tests impairment was defined as performance that was 1.33 SDs below the mean of a reference group of healthy peers. Raw scores indicating impaired performance could be > or < than the mean depending on the test (eg. on tests of accuracy the cut-off will be a score 1.33 SDs below the mean, while on a timed test the cut-off will be 1.33 SDs above the mean).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 1853 | 373 | 720 | 760
Participants | 402 | 46 | 134 | 222
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p < 0.0001, ANOVA

11. Secondary Outcome: 6 Month Trail Making Test (TMT) Part B - Impaired
Description: The TMT is a measure of attention, speed, and mental flexibility. Part A requires the individual to draw lines to connect 25 encircled numbers distributed on a page. Part B is similar except the person must alternate between numbers and letters, is more difficult, takes longer to complete. Both sections are timed, the score represents the amount of time required to complete the task, with shorter times indicating better performance.
  Impairment cutoff: > 143.7 (based on the comparison group as a whole and expressed as raw score).
  For all the cognitive tests impairment was defined as performance that was 1.33 SDs below the mean of a reference group of healthy peers. Raw scores indicating impaired performance could be > or < than the mean depending on the test (eg. on tests of accuracy the cut-off will be a score 1.33 SDs below the mean, while on a timed test the cut-off will be 1.33 SDs above the mean).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 1799 | 365 | 702 | 732
Participants | 368 | 46 | 113 | 209
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p < 0.0001, ANOVA

12. Secondary Outcome: 6 Month Cambridge Neuropsychological Test Automated Battery (CANTAB) PAL (Paired Associate Learning Task) - Impaired
Description: CANTAB is a computerized neuropsychological battery examining a range of domains including attention, memory and executive functioning. Using mainly nonverbal stimuli, the test is language- and culture-independent. For CANTAB PAL, the individual must remember 1 to 8 patterns displayed in different positions on the screen. The score is the number of incorrect responses adjusted if necessary for trials that have not been completed. Scores ranged from 0-194 with lower score indicating better performance.
  Impairment cutoff: > 72.3 (based on the comparison group as a whole and expressed as raw score).
  For all the cognitive tests impairment was defined as performance that was 1.33 SDs below the mean of a reference group of healthy peers. Raw scores indicating impaired performance could be > or < than the mean depending on the test (eg. on tests of accuracy the cut-off will be a score 1.33 SDs below the mean, while on a timed test the cut-off will be 1.33 SDs above the mean).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 1546 | 342 | 587 | 617
Participants | 231 | 42 | 72 | 117
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p = 0.637, ANOVA

13. Secondary Outcome: 6 Month Cambridge Neuropsychological Test Automated Battery (CANTAB) RTI (Reaction Time Task) - Impaired
Description: The CANTAB is a computerized neuropsychological battery examining a range of domains including attention, memory and executive functioning. Using mainly nonverbal stimuli, the test is language- and culture-independent. For CANTAB RTI, the individual must respond as quickly as possible to a circle presented at one of 5 positions. The outcome measure is the median time for correct responses (ms).
  Impairment cutoff: > 470.9 (based on the comparison group as a whole and expressed as raw score).
  For all the cognitive tests impairment was defined as performance that was 1.33 SDs below the mean of a reference group of healthy peers. Raw scores indicating impaired performance could be > or < than the mean depending on the test (eg. on tests of accuracy the cut-off will be a score 1.33 SDs below the mean, while on a timed test the cut-off will be 1.33 SDs above the mean).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 1462 | 321 | 542 | 599
Participants | 237 | 38 | 63 | 136
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p < 0.0001, ANOVA

14. Secondary Outcome: 6 Month Cambridge Neuropsychological Test Automated Battery (CANTAB) SWM (Spatial Working Memory Task) - Impaired
Description: The CANTAB is a computerized neuropsychological battery examining a range of domains including attention, memory and executive functioning. Using mainly nonverbal stimuli, the test is language- and culture-independent. For the CANTAB SWM, the participant searches for tokens in boxes on the screen. The between errors measure is the number of times the participant queries a box that has already been searched. Errors ranged from 0 to 151, with lower numbers indicating better performance.
  Impairment cutoff: > 52.0 (based on the comparison group as a whole and expressed as raw score).
  For all the cognitive tests impairment was defined as performance that was 1.33 SDs below the mean of a reference group of healthy peers. Raw scores indicating impaired performance could be > or < than the mean depending on the test (eg. on tests of accuracy the cut-off will be a score 1.33 SDs below the mean, while on a timed test the cut-off will be 1.33 SDs above the mean).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 1483 | 334 | 564 | 585
Participants | 259 | 49 | 81 | 129
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p = 0.480, ANOVA

15. Secondary Outcome: 6 Month Cambridge Neuropsychological Test Automated Battery (CANTAB) RVP (Rapid Visual Information Processing Task) - Impaired
Description: The CANTAB is a computerized neuropsychological battery examining a range of domains including attention, memory and executive functioning. Using mainly nonverbal stimuli, the test is language- and culture-independent. For the CANTAB RVP, sequences of numbers must be detected as they appear on the screen. The measure of accuracy is A' (A prime) which is derived from hits and correct rejections. The maximum score is 1 and, a higher A' indicates better performance.
  Impairment cutoff: < 0.82 (based on the comparison group as a whole and expressed as raw score).
  For all the cognitive tests impairment was defined as performance that was 1.33 SDs below the mean of a reference group of healthy peers. Raw scores indicating impaired performance could be > or < than the mean depending on the test (eg. on tests of accuracy the cut-off will be a score 1.33 SDs below the mean, while on a timed test the cut-off will be 1.33 SDs above the mean).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 1368 | 311 | 514 | 543
Participants | 225 | 33 | 46 | 146
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p < 0.0001, ANOVA

16. Secondary Outcome: 6 Month Cambridge Neuropsychological Test Automated Battery (CANTAB) SOC (Stockings of Cambridge Task) - Impaired
Description: The CANTAB is a computerized neuropsychological battery examining a range of domains including attention, memory and executive functioning. Using mainly nonverbal stimuli, the test is language- and culture-independent. For the CANTAB SOC, the individual moves circles to match a target in this task based on the Tower of Hanoi game. The score is the number of problems solved in the minimum number of moves, with a maximum of 12. Higher scores indicate better performance.
  Impairment cutoff: < 5.7(based on the comparison group as a whole and expressed as raw score).
  For all the cognitive tests impairment was defined as performance that was 1.33 SDs below the mean of a reference group of healthy peers. Raw scores indicating impaired performance could be > or < than the mean depending on the test (eg. on tests of accuracy the cut-off will be a score 1.33 SDs below the mean, while on a timed test the cut-off will be 1.33 SDs above the mean).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 1440 | 329 | 548 | 563
Participants | 182 | 28 | 64 | 90
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p = 0.024, ANOVA

17. Secondary Outcome: 6 Month Cambridge Neuropsychological Test Automated Battery (CANTAB) AST (Attention Switching Task ) - Impaired
Description: The CANTAB is a computerized neuropsychological battery examining a range of domains including attention, memory and executive functioning. Using mainly nonverbal stimuli, the test is language- and culture-independent. For the CANTAB AST, participants respond either to the position of an arrow or the direction it is pointing, after being cued to the task on each trial. Total correct responses range from 0 to 160, where higher numbers indicate better performance.
  Impairment cutoff: <135.5 (based on the comparison group as a whole and expressed as raw score).
  For all the cognitive tests impairment was defined as performance that was 1.33 SDs below the mean of a reference group of healthy peers. Raw scores indicating impaired performance could be > or < than the mean depending on the test (eg. on tests of accuracy the cut-off will be a score 1.33 SDs below the mean, while on a timed test the cut-off will be 1.33 SDs above the mean).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 1488 | 332 | 559 | 597
Participants | 282 | 49 | 85 | 148
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p = 0.064, ANOVA

18. Secondary Outcome: Early (2-3 Weeks) MRI Imaging - Traumatic Intracranial Abnormalities
Description: A selected number of sites performed MRI follow up in a subset of patients that consented for imaging data collection. The CENTER-TBI MR protocols included a high-resolution 3D T1-weighted, a T2-weighted, a FLAIR, a DTI, a T2* sequence (gradient echo and/or SWI), and (optionally) a resting-state fMRI. Across all stratum the MRI sites performed a follow up MRI at 2-3 weeks after injury.
  Traumatic Intracranial Abnormalities were assessed according to the TBI-Common Data Elements (CDEs). It indicates whether any of the 12 following imaging abnormalities are present (Mass lesion, Extra-axial Hematoma, Epidural Hematoma, Subdural Hematoma Acute, Subdural Hematoma Subacute Chronic, Subdural Collection Mixed Density, Contusion, TAI, traumatic Subarachnoid Hemorrhage, Intraventricular Hemorrhage, Midline Shift or Cisternal Compression.
Time Frame: Between 2-3 weeks after enrolment
Measure: Count of Participants; unit: Participants
Arm/Group | CENTER-TBI Population | ER Stratum | Admission Stratum | ICU Stratum
Number analyzed (Participants) | 504 | 123 | 180 | 197
Participants | 312 | 32 | 101 | 179
Statistical Analysis 1: Comparison: CENTER-TBI Population; null hypothesis: no difference between ER stratum, Admission stratum and ICU stratum; Test type: Non-Inferiority — non-inferiority margin = 0; p < 0.0001, ANOVA

ADVERSE EVENTS:
Time Frame: 2 years
Description: Observational study: no adverse events to be reported since there is no intervention.
  The number of patients admitted to the ICU is seen as the population at risk for all-cause mortality, due to the severity of ICU patients: 2138 patients.
Arm/Group | CENTER-TBI Population
All-Cause Mortality (participants affected / at risk) | 363/2138
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT02210221/Prot_SAP_000.pdf